CLINICAL TRIAL: NCT07101003
Title: A Comparative Evaluation of the Degree of Pain and MMP-9 Expression Following Instrumentation of Necrotic Pulps With Apical Periodontitis in One or Two Visits: A Randomized Clinical Trial
Brief Title: A Comparative Evaluation of the Degree of Pain and MMP-9 Expression Following Instrumentation of Necrotic Pulps With Apical Periodontitis in One or Two Visits
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Marwa Hisham Mohamed Salah Eldin (Other)
Responsible Party: Sponsor-Investigator, Marwa Hisham Mohamed Salah Eldin, Principal Investigator, Cairo University
Organization: Cairo University (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 14422023517120
Record Dates: First submitted 2025-07-28; First posted 2025-08-03 (Actual); Last update posted 2025-08-03 (Actual); Status verified 2025-07

CONDITIONS: Apical Periodontitis; Necrotic Pulps; Single Rooted Teeth
Keywords: necrotic pulps; root canal system; Enterococcus faecalis (E. faecalis); Microbioogy; pain; bacterial reduction; Matrix metalloproteinases (MMPs)
MeSH Terms: conditions — Periapical Periodontitis; Pain

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Multiple instrumentation (Active Comparator): root canal instrumentation will be done on two visits as a control
  Interventions: Procedure: multiple visit instrumentation
- single instrumentation (Experimental): Root canal instrumentation will be done on one visits
  Interventions: Procedure: single visit instrumentation

INTERVENTIONS:
Procedure: single visit instrumentation — root canal instrumentation will be done on single visit treatment
  Arms: single instrumentation
Procedure: multiple visit instrumentation — root canal treatment will be done on two visits
  Arms: Multiple instrumentation

SUMMARY:
This randomized clinical trial compares postoperative pain and MMP-9 levels after root canal treatment of necrotic teeth with apical periodontitis, using either single-visit or two-visit instrumentation. The primary outcome is pain intensity measured at multiple intervals using a Visual Analogue Scale. The secondary outcome is the periapical expression of MMP-9 assessed via ELISA. The trial aims to determine whether treatment timing impacts inflammation and healing.

DETAILED DESCRIPTION:
This randomized clinical trial is designed as a parallel-group superiority study with an allocation ratio of 1:1. It is conducted at the postgraduate outpatient clinic of the Endodontics Department, Faculty of Dentistry, Cairo University. The target population includes adult patients aged between 18 and 40 years who present with straight, single-canaled permanent teeth diagnosed with necrotic pulp and chronic apical periodontitis. The diagnosis is confirmed using clinical criteria such as a negative response to cold testing, absence of spontaneous pain, and radiographic findings showing periapical radiolucency not exceeding 2×2 mm with a PAI score of 2 or 3. Only systemically healthy individuals (ASA I or II) who have not taken antibiotics or anti-inflammatory drugs in the past month and can comprehend the pain scoring system are included. Patients with acute infections, non-restorable teeth, prior root canal treatment, or significant systemic conditions are excluded.

Eligible patients are randomly assigned into two groups using a computer-generated randomization sequence. Allocation is concealed and handled by the co-supervisor. The experimental group receives single-visit root canal instrumentation, while the control group undergoes a two-visit protocol. In both groups, treatment begins with standard diagnostic procedures, local anesthesia, rubber dam isolation, and access cavity preparation. Before instrumentation, a baseline periapical fluid sample (PS-1) is collected by inserting sterile paper points beyond the apex into the canal for 60 seconds and storing them at -80°C for later MMP-9 analysis via ELISA.

In the single-visit group, biomechanical preparation is completed in one session using Fanta Blue rotary files with a 4% taper, progressing to size 40. Irrigation is performed with 2.5% sodium hypochlorite after each file, followed by saline as a final rinse. The access cavity is sealed temporarily with glass ionomer or IRM. Patients are instructed to record postoperative pain using a modified Visual Analogue Scale (VAS) at 6, 12, 24, 48, and 72 hours. One week later, a second periapical sample (PS-2) is collected under local anesthesia and rubber dam isolation.

The control group undergoes a two-visit protocol. In the first visit, canal preparation is only performed up to size 25, with the same irrigation and temporary sealing as in the experimental group. The second visit, one week later, includes collection of the second periapical sample (PS-2), followed by completion of instrumentation to size 40. All patients receive postoperative instructions and pain charts, and are asked to return after three days for chart collection and assessment.

The primary outcome of the study is the intensity of postoperative pain, measured at five time points using the modified VAS. The secondary outcome is the level of MMP-9 expression in the periapical tissues before and after treatment. Data are analyzed using IBM SPSS v22. Normality of data is tested using the Kolmogorov-Smirnov and Shapiro-Wilk tests. If data are normally distributed, independent t-tests are used to compare groups; otherwise, the Mann-Whitney U test is applied. Statistical significance is set at p ≤ 0.05.

To ensure data integrity, all forms are coded, stored securely, and access is restricted to the study team. Blinding is applied to patients, the outcome assessor, the lab technician performing ELISA, and the statistician. The sample size is calculated based on prior literature to detect a clinically significant difference in pain scores, leading to a total enrollment of 28 patients (14 per group), accounting for a 25% dropout rate.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18-40 years.
* Males/Females.
* Straight single canaled permanent teeth:

  * Non-Vital pulps.
  * Negative response to cold pulp tester (ethyl chloride spray*).
  * Absence of spontaneous pain.
  * Chronic apical periodontitis with negative response to percussion
  * Slight widening in the periodontal membrane space or with periapical radiolucency not exceeding 2*2 mm radiographically. The Periapical Index (PAI) score by Ørstavik is 2 or 3 (Ørstavik et al., 1986 43)
* Systemically healthy patients (ASA I or II)
* No anti-inflammatory or antibiotic medications taken in the past month
* Patients' acceptance to participate in the trial.
* Patients who can understand pain scale and can sign the informed consent (Appendix I).
* Patients' acceptance to participate in the trial.

Exclusion Criteria:

* Medically compromised patients having significant systemic disorders. (ASA III or IV).
* Teeth with swelling or fistulous tract.
* Teeth with acute or chronic periapical abscess.
* Mobility Grade II or III.
* Previous root canal therapy.
* Non-restorable teeth.
* Immature teeth.
* Pregnant females.

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 28 (Estimated)
Dates: Start 2025-08-01 (Estimated); Primary Completion 2025-08-01 (Estimated); Study Completion 2025-08-04 (Estimated)

PRIMARY OUTCOMES:
Post instrumentation Pain | At 6,12, 24, 48 and 72 hours post instrumentation
  Pain will be measured At 6,12, 24, 48 and 72 hours post instrumentation by Modified Visual Analogue Scale (VAS)

SECONDARY OUTCOMES:
MMP-9 level | pre-instrumentation & 1 week post-instrumentation
  measure expression of MMP-9 After access cavity (pre-instrumentation & 1 week post-instrumentation

IPD SHARING:
Plan to Share IPD: No